CLINICAL TRIAL: NCT03061565
Title: Long Term Effects of Erythropoietin in Patients With Moderate to Severe Traumatic Brain Injury A Follow-up Study of an International Randomised Controlled Trial
Brief Title: Long Term Effects of Erythropoietin in Patients With Moderate to Severe Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, David James Cooper, Director, Australian and New Zealand Intensive Care Research Centre
Other Study IDs: ANZIC-RC EPO-TBI Long term
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Traumatic Brain Injury
Keywords: erythropoietin; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Erythropoietin; Epoetin Alfa; Sodium Chloride

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Erythropoietin: Patients were treated with EPO during the EPO-TBI study in 2010-2014.
  Interventions: Drug: erythropoietin
- Placebo: Patients were treated with placebo during the EPO-TBI study in 2010-2014.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: erythropoietin — Patients were given erythropoietin during the EPO-TBI study in 2010-2014. In the current follow-up we will evaluate any possible long term differences between patients treated with etrythropoietin compared to placebo.
  Other Names: EPOETIN ALFA
  Groups: Erythropoietin
Drug: Placebos — Patients were given placebo during the EPO-TBI study in 2010-2014. In the current follow-up we will evaluate any possible long term differences between patients treated with etrythropoietin compared to placebo.
  Other Names: Sodium chloride
  Groups: Placebo

SUMMARY:
Traumatic brain injury is catastrophic event that commonly require treatment in an intensive care unit. Management is mainly supportive aiming at avoiding hypoxia, hypotension, hypoglycaemia and increased intracerebral pressure. Thus far efforts to find a specific pharmacologic therapies have been disappointing. Recently it was demonstrated that recombinant erythropoietin has been found to decrease mortality at six months from injury but without significantly improving functional neurological outcome (GOSe). Whether this survival benefit of EPO is sustained beyond 6 months is unknown.

In the current study survival data will be collected centrally and patients alive or person responsible will be invited to participate in an evaluation of neurological function and quality of life. Factors associated with time to death as well as factors associated with long term quality of life will be determined with statistical methods.

DETAILED DESCRIPTION:
Aim: In this post hoc study of a RCT the primary aim is to determine the effect of EPO compared to placebo in improving outcome, including survival, neurological function and quality of life two years after the conclusion of the EPO-TBI study (two to seven years after moderate or severe TBI occurring in individual patients).

Design: A long term follow-up study of a prospective, multi-centre, double blind, phase III, randomised controlled trial.

Methods: Survival status at the time when this follow-up trial is executed will obtained in all patients. Time from injury will vary between 2 to 7 years depending on when the patient was enrolled. This information will obtained from hospital notes, national register offices and/or national statistical bureaus. Since the trial was an international RCT, strategies may vary and will take into account local circumstances. Local plans will be developed by the local principal investigators and approved by the management committee.

Data includes

* Survival status at long term follow up (alive/dead)
* Time from injury to assessment (days)
* If the patients is deceased, time of death and time from injury in days

Quality of life assessment

Patients (or a proxy - generally a close family member) who are alive at 2-7 years after randomisation will be interviewed by trained assessors. The same contact person as used in the primary trial will be contacted primarily. Consent will be obtained for the conduction for long term assessment. Assessors will use a standardized structured telephone questionnaires to determine GOSE and QOL. Neurological outcomes will then be defined as favourable (GOSE 5 to 8; moderate disability and good recovery) or unfavourable (GOSE 1 to 4; death and severe disability). Data include:

* Time of assessment
* Time from injury in days
* Follow-up GOSE
* Follow-up EQ-5D
* Follow-up SF-12

ELIGIBILITY:
Inclusion Criteria:

* Participation in the EPO-TBI study without withdrawal of informed consent.

Exclusion criteria:

* Failure to to consent for the conduction of the follow-up assessment.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The EPO-TBI study conducted between 2010 and 2015 enrolled a total of 606 patients treated for moderate to severe traumatic brain injury in the intensive care unit. Of these consent was withdrawn in 3 patients. Of the 603 patients, 524 we alive at 6 months. Survival status will be checked in these 524 patients and those alive will be included in a follow-up of functional recover and quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality and time to mortality at least 2 years from injury | 2-7 years from injury
  Survival status with time to death in those deceased

SECONDARY OUTCOMES:
Glasgow outcome scale extended | 2-7 years from injury
  Neurological outcome
SF-12 | 2-7 years from injury
  Quality of life scale
EQ-5D | 2-7 years from injury
  Quality of life scale

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo Bellomo, Principal Investigator — ANZIC-RC Monash University
Locations (1):
- Australian and New Zealand Intensive Care Research Centre, Monash University, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No